CLINICAL TRIAL: NCT00357734
Title: Multicenter Open-label, Long-term Safety Trial of Treatment Extension With ZD1839 in Patients Who Have Been Treated in Other ZD1839 Clinical Trials.
Brief Title: Iressa Follow-up Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0555; D7913L00008
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer; Breast Cancer
Keywords: lung cancer; breast cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefitinib (ZD1839) (Experimental): ZD1839 at a daily dose of 250 mg or 500 mg depending on final dose in parent trial
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — ZD1839 at a daily dose of 250 mg or 500 mg depending on final dose in parent trial

SUMMARY:
The purpose of this study is to assess the long-term safety profile and the secondary objective to estimate clinical benefit of ZD1839 (gefitinib).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent to participate in the trial.
* Female or male aged 18 years and over.
* Patients with previously diagnosed cancer who have been treated with ZD1839 in a parent ZD1839 clinical trial and may benefit from continuation

Exclusion Criteria:

* Known severe hypersensitivity to ZD1839
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort.
* Withdrawal from a parent ZD1839 trial because of tumor progress

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Germany Medical Director, MD, Study Director — AstraZeneca
Locations (7):
- Germany (7):
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Großhansdorf
  - Research Site, Hemer
  - Research Site, Jena
  - Research Site, Minden
  - Research Site, Tübingen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 16 June 2005, Last subject last visit: 18 May 2015. The study was conducted in Germany.
Period: Overall Study
Arm/Group | Gefitinib (ZD1839)
Started | 14
Patients Received 250 mg of ZD1839 | 13
Patient Received 500 mg of ZD1839 | 1
Completed | 10
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Gefitinib (ZD1839)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: Years] | 66 [52 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4

OUTCOME MEASURES:

1. Secondary Outcome: Progression-free Survival (PFS)
Description: Objective disease progressing was assessed using the previous cancer response criteria in the parent ZD1839 trial: ie Southwest Oncology Group (SWOG) tumor response criteria, as a 50% increase or an increase of 10 cm2 (whichever is smaller) in the sum of products of all measurable lesions from the overall smallest sum observed (over baseline if no decrease) using the same techniques as baseline; Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase In the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From randomization until progression or death (up to 120 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib (ZD1839)
Number analyzed (Participants) | 14
Months | 26.5 [11 to 56]

2. Secondary Outcome: Overall Survival (OS)
Time Frame: From randomization until death (up to 120 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib (ZD1839)
Number analyzed (Participants) | 14
Months | 23.5 [15 to 56]

3. Primary Outcome: Number of Serious Adverse Events (SAEs)
Description: Assessment of the long-term safety profile of ZD1839 therapy by assessing the incidence of adverse events. Any adverse events (AEs) and serious adverse events (SAEs) occurring during treatment and any SAEs occurring within 30 days after stopping the trial drug must be followed to resolution unless, in the investigator's opinion, the condition is unlikely to resolve because of the patient's underlying disease
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment until 30 days after the last dose of study treatment or 30 days after last visit (up to approximately 120 months)
Measure: Number; unit: number of SAEs
Arm/Group | Gefitinib (ZD1839)
Number analyzed (Participants) | 14
number of SAEs | 13

4. Primary Outcome: Number of Serious Adverse Events (SAEs) Related to ZD1839
Description: as for outcome 3
Time Frame: as for outcome 3
Measure: Number; unit: Number of SAEs related to ZD1839
Arm/Group | Gefitinib (ZD1839)
Number analyzed (Participants) | 14
Number of SAEs related to ZD1839 | 0

5. Primary Outcome: Number of Other Adverse Events (AEs)
Description: as for outcome 3
Time Frame: as for outcome 3
Measure: Number; unit: number of other AEs
Arm/Group | Gefitinib (ZD1839)
Number analyzed (Participants) | 14
number of other AEs | 40

6. Primary Outcome: Number of Other Adverse Events (AEs) Related to ZD1839
Description: as for outcome 3
Time Frame: as for outcome 3
Measure: Number; unit: number of other AEs related to ZD1839
Arm/Group | Gefitinib (ZD1839)
Number analyzed (Participants) | 14
number of other AEs related to ZD1839 | 19

ADVERSE EVENTS:
Arm/Group | Gefitinib (ZD1839)
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (ZD1839) (N=14)
Duodenitis (Gastrointestinal disorders) | 1 — Causality to study medication: No
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 — Causality to study medication: No
Vomiting (Gastrointestinal disorders) | 1 — Causality to study medication: No
Ascites (Gastrointestinal disorders) | 1 — Causality to study medication: No
Bronchopneumonia (Infections and infestations) | 1 — Causality to study medication: No
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 — Causality to study medication: No
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 — Causality to study medication: No
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Causality to study medication: No
Death (General disorders) | 1 — Causality to study medication: No
Asthenia (General disorders) | 1 — Causality to study medication: No
Haematemesis (Gastrointestinal disorders) | 1 — Causality to study medication: No
General physical health deterioration (General disorders) | 1 — Causality to study medication: No
Pneumonia (Infections and infestations) | 1 — Causality to study medication: No
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (ZD1839) (N=14)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
DIZZINESS (Nervous system disorders) | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
ANAEMIA (Blood and lymphatic system disorders) | 1
COLITIS (Gastrointestinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
EPIDIDYMITIS (Infections and infestations) | 1
FATIGUE (General disorders) | 1
GALLBLADDER PAIN (Hepatobiliary disorders) | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
NAUSEA (Gastrointestinal disorders) | 3
OEDEMA (General disorders) | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1
PARONYCHIA (Infections and infestations) | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 3
WEIGHT DECREASED (Investigations) | 1
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The study was stopped after enrolling 14 of 100 patients. The outcome was biased by the limited number of patients. Therefore, data allow only a limited statement on efficacy and long term safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less